CLINICAL TRIAL: NCT01690910
Title: Effects of Mobility Devices on Nursing Compliance With Mobility Protocols.
Acronym: EMS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Patient enrollment to low to support an analysis
Sponsor: Trinity Health Michigan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RCAY 40
Record Dates: First submitted 2012-08-31; First posted 2012-09-24 (Estimated); Results first posted 2021-04-13 (Actual); Last update posted 2021-04-13 (Actual); Status verified 2021-03

CONDITIONS: Mobility Limitations
Keywords: Ventilator; Mobility Limitations; Critical Care; Rifton Gait Trainer
MeSH Terms: conditions — Mobility Limitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Front Wheeled Walker (Active Comparator): The Front Wheeled Walker is a standard walker that is used to assist patients while walking.
  Interventions: Device: Front Wheeled Walker
- Rifton Gait Trainer (Active Comparator): The Rifton Gait Trainer is used to assist patients while walking. It includes a harness to support the patient and prevent falls.
  Interventions: Device: Rifton Gait Trainer

INTERVENTIONS:
Device: Rifton Gait Trainer
  Arms: Rifton Gait Trainer
Device: Front Wheeled Walker
  Arms: Front Wheeled Walker

SUMMARY:
This is a 10-week pilot study for a randomized non-blinded controlled clinical trial to assess whether use of the Rifton Gait Trainer will improve the incidence of mobilization of critically ill ventilator dependent patients in the intensive care units (ICUs) and improve important patient outcomes. The pilot study is designed to assess the feasibility and logistics of doing a study of this nature in the ICU; it will also provide the means to obtain estimates of outcome effect sizes, number of repeated measures, time between repeated measures, and intra-subject and intra-unit correlations, to be used for sample size calculations.

DETAILED DESCRIPTION:
Background Critical care costs an estimated 90 billion dollars per year in the United States, comprising approximately 1% of the gross national product.1 Though this expenditure is enormous, together with advances in critical care medicine and mechanical ventilation technology, it has produced a priceless trend in decreasing intensive care unit (ICU) mortality.1 Of all ICU admissions, about 40% require mechanical ventilation, often with accompanying necessary periods of sedation and inactivity.1 Although more patients are surviving their ICU stay, it is becoming apparent that our current ICU culture of heavy sedation and inactivity is taking its toll on the complete recovery of the critically ill patient. 1,2 Several studies have shown significant disability one year after discharge, as well as major declines in functional status and health-related quality of life; half of ICU patients were unable to return to work due to persistent fatigue, weakness, and poor functional status. 4 The primary contributor was muscle wasting and weakness,5 due to the prolonged immobilization brought about by illness, lengthy bed rest, deep sedation, and the use of paralytic agents.6 It is estimated that just a single day of inactivity causes muscle strength to decrease by 1-1.5%.7 Although 94% of survivors with critical illness myoneuropathy can demonstrate meaningful clinical recovery of muscle strength 9 months out from their hospital stay, there are still some patients whose weakness may persist, resulting in severe and prolonged functional deficits.14,18 To combat the deleterious effects of inactivity and improve complete recovery, some hospitals have instituted programs under the rubric early mobility, wherein sedation is reduced and patients are engaged in progressive levels of activity as soon as physically possible. Early mobilization starts with passive range of motion exercises, then progresses to active range of motion, sitting, standing, and, finally, walking. Early mobility in the ICU has been proposed as a crucial instrument in muscle preservation and protection from neuropathy of critical illness, thereby decreasing long-term morbidity and physical debilitation.18

There is a growing body of evidence indicating that early mobilization of ventilated patients can have a significant positive impact on length of stay, muscle condition, and the patient's overall sense of well-being. The use of early mobility in patients with respiratory failure has been proven safe with the implementation of proper monitoring in a physiologically stable and awake patient.2 Hopkins et al. implemented an early activity program and demonstrated a decline in length of ICU stay of 3 days.1 Morris et al. implemented a similar early mobilization program that showed a statistically significant decrease in the length of stay in the ICU (6.9 vs. 5.5 days, P=0.025) as well as in the hospital (14.5 vs. 11.2 days, P=0.006); in addition there was a notable trend towards decreased inpatient cost per patient ($44,302 vs. $41,142, P=0.262).19 Schweikert et al. were able to demonstrate that patients who had undergone early mobilization had a greater rate of return to independent functional status at hospital discharge (59% vs. 35%, P=0.02).20 These studies have demonstrated the ability to increase mobilization, improve physical function, and decrease ICU resource utilization within a relatively short period of time with an appropriate change in routine clinical practice.12

Unfortunately, there exist significant barriers to the implementation of an early mobility program. The most significant and pervasive of these barriers is cultural-the perception that the critically ill patient cannot tolerate physical activity. This barrier, however, is rapidly dissolving with the mounting evidence noted above. The demonstrated benefits of early mobility have prompted increasing numbers of institutions to develop their own early mobility protocols and attempt their implementation. Once the cultural barriers are overcome, however, additional barriers appear. Thus, implementation has been slow and spotty. In a multisite study, only 27% of patients with acute lung injury received any form of physical therapy in the ICU, with treatments occurring only 6% of those days.22 These barriers involved: 1) providing safety guarantees, 2) accommodating staffing models, and 3) finding the right hardware. With regard to safety guarantees, there exist legitimate fears regarding possible harm to the patient in the process of mobilization, either secondary to patient falls, or unintentional removal of lines, feeding or drainage tubes, or endotracheal tubes. Safe mechanical support is needed for the patient, to the point of full body-weight support. The staffing model is also critical: the mobilization of one ventilated patient requires, in addition to a physical therapist, at least three staff members to move medical equipment while the patient walks.11, 21 Although on a given day, within a 20-bed ICU, only two patients might qualify for assisted walking, and would require only four 15-minute periods from a 5-member mobility team per day, the logistics of assembling that team from the ICU staff are often prohibitive. Finally with regard to finding appropriate hardware, the management and transport of medical equipment alongside the walking patient is not easily addressed with rolling poles and carts. The current standard of care for walking a mechanically ventilated patient consists of a wheeled walker held onto by the patient, the patient supported with a gait belt held from behind by a physical therapist, and 4-5 staff persons in attendance to guide the patient, roll the equipment, and be ready to "pick up" should the patient fall.

As an alternative to the front-wheeled walker, the Rifton Gait Trainer has been introduced into clinical practice. This device provides greater inherent safety features via a pelvic harness that keeps the patient from falling, even if their legs should give out while walking. In addition, there is a chest piece to keep patients from tipping forward or backward, and there are higher handholds to help patients mobilize more easily. The Rifton Gait Trainer addresses two of the three above listed barriers by providing more inherent safety features through better hardware, and it may also help decrease the number of staff required to mobilize patients.

Purpose The following sections describe a 10-week pilot study for a randomized non-blinded controlled clinical trial to assess whether use of the Rifton Gait Trainer will improve the incidence of mobilization of critically ill ventilator dependent patients in the intensive care units (ICUs) and improve important patient outcomes. The pilot study is designed to assess the feasibility and logistics of doing a study of this nature in the ICU; it will also provide the means to obtain estimates of outcome effect sizes, number of repeated measures, time between repeated measures, and intra-subject and intra-unit correlations, to be used for sample size calculations for a multi-center study.

Subjects Approximately forty subjects will be randomized to use either the RGT or the FWW, with enrollment spanning a period of approximately 10 weeks. Patients will be deemed eligible to ambulate based on their daily mobility score, as calculated according to the Early Mobility Protocol. Mobility scores are first determined based on level of consciousness. The unconscious patient has the lowest mobility level, Level 1. Patients who are conscious but have a low RASS score (-2) are considered a Level 2. Conscious patients are considered to be Level 3 or 4. Level 4 patients are those patients who have proven that they can master all the activities outlined for Level 3 mobility; that is, they can dangle at the bedside and stand and pivot to a chair. Level 4 activities are separated from Level 3 activities only by the ability to walk in the hallway.

Informed consent will occur prior to randomization. Randomization will occur when patients have been on the ventilator > 2 days and have mobility scores eligible for walking. Randomization will be assigned on a 1:1 ratio to either the RGT or FWW. Patients will be randomized using a web-based system called CREDIT.

Data Analysis A future study will be considered feasible if we are able to enroll 60% of eligible patients, have records for 90% of eligible ambulation days, and at least 85% of required data fields are completed as designed. Analysis will be based on intention-to-treat; that is, regardless of which walker is actually used, the patient will be analyzed in the group to which he or she was randomized.

The primary outcome measure, how many times the patient is mobilized each day, will be compared between devices using a hierarchical generalized linear model with number of times the patient is mobilized each day as the dependent variable, device, unit and day and an interaction of device with day as the independent variables, and subject as the random effect in the model. Most likely, ordinal regression will be used with 0, 1, 2 or more times as the definition of outcome. If there are too few occurrences of 2 or more, we will convert to a logistic model. If one device is better than the other, we would expect the odds of being mobilized at a higher level with RGT is significantly different from the odds of being mobilized with FWW. We will also test for the interaction of device with time.

Sources

ELIGIBILITY:
Inclusion Criteria:

* >18 years of age
* On the ventilator for > 48 hours
* Mobility score > 3

Exclusion Criteria:

* > 220 lbs
* Limb amputees
* Prisoners
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2012-09; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MaryAnne Purtill, MD, Principal Investigator — St. Jospeh Mercy Hospital
Locations (1):
- Saint Joseph Mercy Hospital, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hopkins RO, Spuhler VJ, Thomsen GE. Transforming ICU culture to facilitate early mobility. Crit Care Clin. 2007 Jan;23(1):81-96. doi: 10.1016/j.ccc.2006.11.004. PMID 17307118
- [Background] Bailey P, Thomsen GE, Spuhler VJ, Blair R, Jewkes J, Bezdjian L, Veale K, Rodriquez L, Hopkins RO. Early activity is feasible and safe in respiratory failure patients. Crit Care Med. 2007 Jan;35(1):139-45. doi: 10.1097/01.CCM.0000251130.69568.87. PMID 17133183
- [Background] Herridge MS, Cheung AM, Tansey CM, Matte-Martyn A, Diaz-Granados N, Al-Saidi F, Cooper AB, Guest CB, Mazer CD, Mehta S, Stewart TE, Barr A, Cook D, Slutsky AS; Canadian Critical Care Trials Group. One-year outcomes in survivors of the acute respiratory distress syndrome. N Engl J Med. 2003 Feb 20;348(8):683-93. doi: 10.1056/NEJMoa022450. PMID 12594312
- [Background] Needham DM, Korupolu R, Zanni JM, Pradhan P, Colantuoni E, Palmer JB, Brower RG, Fan E. Early physical medicine and rehabilitation for patients with acute respiratory failure: a quality improvement project. Arch Phys Med Rehabil. 2010 Apr;91(4):536-42. doi: 10.1016/j.apmr.2010.01.002. PMID 20382284
- [Background] Fan E, Zanni JM, Dennison CR, Lepre SJ, Needham DM. Critical illness neuromyopathy and muscle weakness in patients in the intensive care unit. AACN Adv Crit Care. 2009 Jul-Sep;20(3):243-53. doi: 10.1097/NCI.0b013e3181ac2551. PMID 19638746
- [Background] Needham DM. Mobilizing patients in the intensive care unit: improving neuromuscular weakness and physical function. JAMA. 2008 Oct 8;300(14):1685-90. doi: 10.1001/jama.300.14.1685. PMID 18840842
- [Background] Morris PE, Goad A, Thompson C, Taylor K, Harry B, Passmore L, Ross A, Anderson L, Baker S, Sanchez M, Penley L, Howard A, Dixon L, Leach S, Small R, Hite RD, Haponik E. Early intensive care unit mobility therapy in the treatment of acute respiratory failure. Crit Care Med. 2008 Aug;36(8):2238-43. doi: 10.1097/CCM.0b013e318180b90e. PMID 18596631
- [Background] Schweickert WD, Pohlman MC, Pohlman AS, Nigos C, Pawlik AJ, Esbrook CL, Spears L, Miller M, Franczyk M, Deprizio D, Schmidt GA, Bowman A, Barr R, McCallister KE, Hall JB, Kress JP. Early physical and occupational therapy in mechanically ventilated, critically ill patients: a randomised controlled trial. Lancet. 2009 May 30;373(9678):1874-82. doi: 10.1016/S0140-6736(09)60658-9. Epub 2009 May 14. PMID 19446324
- [Background] Needham DM, Wang W, Desai SV, Mendez-Tellez PA, Dennison CR, Sevransky J, Shanholtz C, Ciesla N, Spillman K, Pronovost PJ. Intensive care unit exposures for long-term outcomes research: development and description of exposures for 150 patients with acute lung injury. J Crit Care. 2007 Dec;22(4):275-84. doi: 10.1016/j.jcrc.2007.02.001. Epub 2007 Jun 27. PMID 18086397

RESULTS

PARTICIPANT FLOW:
Groups:
- Front Wheeled Walker: The Front Wheeled Walker is a standard walker that is used to assist patients while walking.
  Front Wheeled Walker
- Rifton Gait Trainer: The Rifton Gait Trainer is used to assist patients while walking. It includes a harness to support the patient and prevent falls.
  Rifton Gait Trainer
Period: Overall Study
Arm/Group | Front Wheeled Walker | Rifton Gait Trainer
Started | 0 (The study was never completed due to feasibility issues.) | 0
Completed | 0 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The study was never completed due to feasibility issues.
Groups:
- Total: Total of all reporting groups
Arm/Group | Front Wheeled Walker | Rifton Gait Trainer | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Continuous
Sex: Female, Male

OUTCOME MEASURES:

1. Primary Outcome: Total Number of Times the Critically Ill Ventilator Dependent Patient is Mobilized.
Time Frame: Duration of Intensive Care Unit Stay (2-30 days)
Population: The study was never completed due to feasibility issues.
Arm/Group | Front Wheeled Walker | Rifton Gait Trainer
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Length of Time the Critically Ill Ventilator Dependent Patient is Mobilized.
Time Frame: Patient weight baring to patient seated (1-12 minutes)
Population: The study was never completed due to feasibility issues.
Arm/Group | Front Wheeled Walker | Rifton Gait Trainer
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Not applicable; study was never started
Arm/Group | Front Wheeled Walker | Rifton Gait Trainer
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No